CLINICAL TRIAL: NCT05947513
Title: Feasibility, Safety, and Efficacy of Concomitant Curcumin in Patients Undergoing Palliative Radiotherapy for FIGO Stage IIIB-IVA Cervical Cancer: An Open-label Pilot Trial
Brief Title: Concomitant Curcumin Palliative Radiotherapy in Advanced Cervical Cancer Trial
Acronym: CuPRAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Addis Ababa University (Other)
Collaborators: Akay Natural Ingredients Private Limited (Unknown)
Responsible Party: Principal Investigator, Biniyam Girma, Principal Investigator, Addis Ababa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001/21/SoP
Record Dates: First submitted 2023-06-21; First posted 2023-07-17 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Cervical Cancer
Keywords: Curcumin; Cervical cancer; Radiosensitizer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concurrent Curcumin Palliative Radiotherapy (Experimental): Daily 1000 mg oral CGM Curcumin in four divided doses for seven days prior to the start of and for three to five weeks concurrently with palliative radiotherapy.
  Interventions: Drug: Curcumin; Radiation: Palliative radiotherapy

INTERVENTIONS:
Drug: Curcumin — Curcumin formulation with enhanced bioavailability which contains food-grade curcumin 35% (w/w) combined with the galactomannan fiber from fenugreek seeds.
  Other Names: Curcumagalactomannoside (CGM); CurQfen
Radiation: Palliative radiotherapy — As per the treatment guidelines of the Tikur Anbessa Hospital Radiotherapy Center, standard-of-care palliative or non-radical radiotherapy entails treatment of advanced cervical cancer patients at a biologically effective dose of 45-55 Gy over the course of three to five weeks.
  Other Names: Non-radical radiotherapy

SUMMARY:
The goal of this clinical trial is to test curcumin as an adjunct treatment in patients with cervical cancer receiving standard-of-care palliative radiation. The main questions it aims to answer are:

1. Is adding curcumin to standard-of-care palliative radiotherapy of cervical cancer patients feasible? Is conducting this study feasible?
2. Does adding curcumin to standard-of-care palliative radiotherapy of cervical cancer patients improve therapeutic responses?
3. Is adding curcumin to standard-of-care palliative radiotherapy of cervical cancer patients safe?
4. How much curcumin is absorbed into the body and how long will it stay in the body?

Participants will:

i. Take 250 mg curcumin capsules four times per day for 4-6 weeks in addition to the prescribed palliative radiotherapy.

ii. Provide blood and urine samples for laboratory tests. iii. Provide blood samples to measure curcumin levels in their body. iv. Obtain CT-scan to measure their tumor response. v. Complete questioners to measure improvements to their quality of life, if any.

ELIGIBILITY:
Inclusion criteria:

* Age >18 years old (Adult, Older Adult)
* Histologically confirmed squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma of the cervix, FIGO stage IIIB-IVA
* Undergoing for standard of care palliative radiotherapy without chemotherapy as per the local treatment guideline
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, 2
* Adequate liver function (aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN (Upper Limit of Normal); total serum bilirubin ≤1.5 x ULN); blood cell counts (absolute neutrophils count ≥1.500/mm3; platelet count ≥100.000/mm3; hemoglobin ≥10.0 g/dL); renal function (serum creatinine ≤1.5 x ULN; estimate creatinine clearance (Cockcroft-Gault) ≥60 mL/min)
* Participants must have measureable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST) V1.1.
* Agree to use an effective form of contraception (e.g., true abstinence (not periodic abstinence), barrier contraception, highly effective hormonal contraception) if the participant is of child bearing age
* Give informed consent

Exclusion criteria:

* Cervical cancer patients who are candidates for single dose palliative radiotherapy
* Patients with severe or bilateral hydronephrosis
* Evidence of distant metastases
* Receiving any other investigational agent concurrently or within the last 4 weeks before enrollment
* Received any previous radiation or chemotherapy for cervical cancer
* Underwent surgery in the four weeks prior to the enrolment date or scheduled to undergo surgery within eight weeks after end of treatment
* Currently using of any chemotherapy or scheduled to receive within eight weeks after end of treatment
* Known allergy to turmeric or its derivatives (ginger, curry, cumin, or cardamom)
* Known allergy to fenugreek, peanut, soy, lentil, pea, bean, and chickpea
* Presence of conditions that precludes the safe administration of the trial intervention and/or prohibit adequate compliance to study requirements including chronic ongoing infections (like HIV, Hepatitis B or C), uncontrolled hypertension, heart failure, cardiac arrhythmia, unstable angina, chronic obstructive lung disease, diabetes mellitus, chronic renal disease, chronic liver disease, biliary tract obstruction or cholelithiasis, gastric or duodenal ulcers, autoimmune or inflammatory disorders, a coagulation or platelet disorder, seizure disorders and psychiatric illness. Patients with disorders other than the ones specified above may also be excluded based on the judgment of the principal investigator.
* Pregnant and breastfeeding women
* Participants with circumstances that will not permit completion of the study or required follow-up. For instance, if travel to and from treatment site is an issue.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Treatment Fidelity Rate | From initiation (Day 1) up to end of treatment over 4-6 weeks
  Proportion of participants who received the study treatment as planned
Objective Response Rate (ORR) | Time Frame: 13-17 weeks
  Objective Response Rate is defined as proportion of participants having a complete response (CR) or partial response (PR) as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) as Assessed by CTCAE v5.0 | Up to 10-14 weeks from treatment initiation
  Any new or worsening of a pre-existing untoward sign, symptom, or disease, including a clinically significant laboratory or vital sign abnormality during study treatment, is defined as a treatment emergent adverse event
Incidence of Dose Reduction in curcumin and radiotherapy regimens | : From initiation (Day 1) up to end treatment over 4-6 weeks
  Incidence of Dose A dose reduction is a decrease in dose from the protocol planned starting dose or a decrease from the previous non-zero dose, even if this decrease has been directly preceded by an interruption in curcumin and radiotherapy regimens
Incidence of Dose Interruption in curcumin and radiotherapy regimens | From initiation (Day 1) up to end treatment over 4-6 weeks
  A Dose Interruption is defined a zero dose given on one or more days on which the protocol-specified dose is non-zero, followed by resumption of dosing
Dose Intensity (DI) of curcumin and radiotherapy | From initiation (Day 1) up to end treatment over 4-6 weeks
  Dose intensity is defined as cumulative dose divided by the treatment duration in weeks
Relative Dose Intensity (RDI) of curcumin and radiotherapy | From initiation (Day 1) up to end treatment over 4-6 weeks
  Relative dose intensity is defined as dose intensity (actual DI) divided by the protocol weekly dose (planned DI), expressed as a percentage.
Disease Control Rate (DCR) | 13-17 weeks
  Disease control rate (DCR): proportion of participants having a complete response (CR) or partial response (PR) or stable disease (SD) as defined by the RECIST 1.1 criteria.
Change from baseline in Health-Related Quality of Life (QOL) as assessed using EORTC QLQ-C30 at 7-9 weeks | Baseline, 7-9 weeks
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) measures quality of life in cancer patients by evaluating physical, psychological, and social functions. Possible scores range from zero to 100, with a higher scale score indicating a higher response level. As such, high scores on functional and global health status (QoL) scales indicate healthy levels of functioning and high quality of life, respectively. However, a high score on the symptoms scale or item indicates more problems or symptomatology.
Change from baseline in Health-Related Quality of Life (QOL) as assessed using EORTC QLQ-C30 at 13-17 weeks | Baseline, 13-17 weeks
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) measures quality of life in cancer patients by evaluating physical, psychological, and social functions. Possible scores range from zero to 100, with a higher scale score indicating a higher response level. As such, high scores on functional and global health status (QoL) scales indicate healthy levels of functioning and high quality of life, respectively. However, a high score on the symptoms scale or item indicates more problems or symptomatology.
Change from baseline in Health-Related Quality of Life (QOL) as assessed using EORTC QLQ-CX24 at 7-9 weeks | Baseline, 7-9 weeks
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Cervical Cancer Module (EORTC QLQ-CX24) measures quality of life in cervical cancer patients in combination with the QLQ-C30. Possible scores range from zero to 100 for all scale and single-item measures. While a high score on the functional single-items indicates a high degree of functioning, a high score on the symptom scales or single-items indicates a high level of symptomatology or difficulties.
Change from baseline in Health-Related Quality of Life (QOL) as assessed using EORTC QLQ-CX24 at 13-17 weeks | Baseline, 13-17 weeks
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Cervical Cancer Module (EORTC QLQ-CX24) measures quality of life in cervical cancer patients in combination with the QLQ-C30. Possible scores range from zero to 100 for all scale and single-item measures. While a high score on the functional single-items indicates a high degree of functioning, a high score on the symptom scales or single-items indicates a high level of symptomatology or difficulties.
Peak Plasma Concentration (Cmax) of CGM Curcumin | Day 1: pre-dose, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours and 6 hours post-dose; Day 6: 30 minutes before the next daily dose, and 1 hour post- dose
  Peak Plasma Concentration represents the highest observed curcumin concentration observed in plasma over all PK sample concentrations following single-dose CGM Curcumin administration.
Time to Peak Plasma Concentration (Tmax) of CGM Curcumin | Day 1: pre-dose, 30 minutes, 1 hour, 1.5 hours, 2hours, 4 hours and 6 hours post-dose; Day 6: 30 minutes before the next daily dose, and 1 hour post- dose
  Time to Peak Plasma Concentration (Tmax) represents the time when Cmax of curcumin occurs following single-dose CGM Curcumin administration.
Area under the Plasma Concentration versus Time Curve (AUCτ) of CGM Curcumin | Day 1: pre-dose, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours and 6 hours post-dose; Day 6: 30 minutes before the next daily dose, and 1 hour post- dose
  Area under the Plasma Concentration versus Time Curve (AUCτ) represents the area under the concentration-time curve of curcumin from time zero to the time of the end of dosing interval following single-dose CGM Curcumin administration.
Half-life (T1/2) of CGM Curcumin | Day 1: pre-dose, 30 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours and 6 hours post-dose; Day 6: 30 minutes before the next daily dose, and 1 hour post- dose
  Half-life (T1/2) represents the time for plasma concentration of curcumin to fall by a factor of one-half in the terminal phase following single-dose CGM Curcumin administration.
Recruitment Rate | through study completion, an average of 1 year
  Recruitment Rate is defined as the proportion of those who participate in the trial who were approached as potential participants.
Assessment Completion Rate | through study completion, an average of 1 year
  Assessment Completion Rate is defined as the proportion of assessments that could be completed as planned.
Attrition Rate | through study completion, an average of 1 year
  Attrition Rate is defined as the proportion of participants who withdraw from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Eyasu Makonnen, Bpharm, PhD, Study Chair — Addis Ababa University; Biniyam Girma, Bpharm, MSc, Study Director — Addis Ababa University; Wondemagegnehu Tigeneh, MD, MMed(RT), Principal Investigator — Addis Ababa University
Locations (1):
- Tikur Anbessa Specialized Hospital, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: No